CLINICAL TRIAL: NCT02211729
Title: A Trial of Seasonal Malaria Chemoprevention Plus Azithromycin in African Children
Acronym: SMCAZ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MR/K007319/1
Record Dates: First submitted 2014-07-17; First posted 2014-08-07 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Malaria; Respiratory Infections
MeSH Terms: conditions — Malaria; Respiratory Tract Infections | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seasonal malaria chemoprevention (Active Comparator): Sulphadoxine-Pyrimethamine Amodiaquine Placebo Azithromycin
  Interventions: Drug: Sulphadoxine-pyrimethamine + amodiaquine + placebo azithromycin
- seasonal malaria chemoprevention plus AZ (Experimental): Sulphadoxine-Pyrimethamine+ Amodiaquine + Azithromycin 4 rounds during malaria transmission season
  Interventions: Drug: Sulphadoxine-Pyrimethamine+ Amodiaquine+ Azithromycin

INTERVENTIONS:
Drug: Sulphadoxine-Pyrimethamine+ Amodiaquine+ Azithromycin — Sulphadoxine-Pyrimethamine+ Amodiaquine+ Azithromycin 4 rounds during malaria transmission season
  Arms: seasonal malaria chemoprevention plus AZ
Drug: Sulphadoxine-pyrimethamine + amodiaquine + placebo azithromycin — Sulphadoxine-pyrimethamine + amodiaquine + placebo azithromycin 4 rounds during malaria transmission season
  Arms: Seasonal malaria chemoprevention

SUMMARY:
The primary objective of this study is to determine whether addition of azithromycin (AZ) to Seasonal Malaria Chemoprevention (SMC) using sulphadoxine/pyrimethamine (SP) +amodiaquine (AQ) will provide an additional reduction in deaths and severe illness in young African children. The secondary objectives include an assessment of the safety and cost-effectiveness of the addition of AZ to SMC with SP+AQ.

This a double blind, randomised, placebo controlled trial. The unit of randomisation will be the household. Children aged 3 - 59 months will be randomised to receive four cycles of either SP+AQ+AZ or SP+AQ+ placebo at monthly intervals during the peak malaria transmission season.

Study Sites: Hounde district in Burkina Faso and in Bougouni district, Mali. Children of 3-59 months of age at the start of each period of drug administration will be eligible for inclusion in the trial provided that parental consent is obtained. Children with a severe, chronic illness or known allergy to one of the study drugs will be excluded.

Primary endpoint: Incidence of the combination of death or hospital admission for at least 24 hours, not due to trauma or elective surgery during the intervention period

Secondary endpoints:

1. incidence of the primary endpoint during the whole study period
2. attendance at a study health centre with a nonmalaria febrile illness
3. attendance at a study health centre with malaria,
4. the prevalence of moderate anaemia at the end of each malaria transmission season,
5. nutritional status at the end of each malaria transmission season,
6. prevalence of nasopharyngeal carriage with pneumococci and macrolide resistant pneumococci before and at the end of each malaria transmissions season,
7. prevalence of resistance markers to SP at the end of the study,

Sample size: 19,200 children (9600 in each country) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex aged 3-59 months of age at the start of each period of drug administration
* parental consent is obtained.

Exclusion Criteria:

* a severe, chronic illness,
* a known allergy to one of the study drugs.
* HIV+ children on cotrimoxazole prophylaxis

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22090 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
severe morbidity and mortality | from the time of enrolment upto the end of malaria transmission in year 3 ( the person time at risk will be restricted to three malaria transmission seasons)
  Incidence of the combination of death or hospital admission for at least 24 hours, not due to trauma or elective surgery during the intervention period.

SECONDARY OUTCOMES:
macrolide resistant pneumococci carriage | before administration of first dose of SMC and at the end of malaria transmission season in year 1, 2 and 3,

OTHER OUTCOMES:
out patient attendance for non malaria febrile illness | from enrolment until the end of malaria transmission season in year 3
  (b) attendance at a study health centre with a febrile illness that is not due to malaria (including acute respiratory infections and diarrhoea),
OPD attendance for malaria | from enrollment until the end of malaria transmission season in year 3
  (c) attendance at a study health centre with RDT or microscopically proven malaria,
moderate anaemia | at the end of each malaria transmission season in year 1, 2, and 3
  (d) the prevalence of moderate anaemia (Hb <8 g/dL) at the end of each malaria transmission season,
nutritional status | at the end of malaria transmission season in year 1, 2 and 3
  (e) nutritional status at the end of each malaria transmission season,
nasopharyngeal carriage | before the administration of first dose of SMC and at the end of malaria transmission season in year 1, 2, and 3
  (f) the prevalence of nasopharyngeal carriage with pneumococci before and at the end of each malaria transmissions season,
SP resistance markers | at the end of the malaria transmission season in year 3
  (h) the prevalence of resistance markers to SP in children with Plasmodium falciparum malaria at the end of the study,
adverse events | 7 days after administration of SMC in rounds 1, 2, 3 and 4 in year one
  solicited adverse events 7 days after administration of SMC+AZ after each round in the year one of the study

CONTACTS AND LOCATIONS:
Locations (2):
- Hounde district Hospital, Houndé, Burkina Faso
- Bougouni Koulikoro District hospital, Bougouni, Mali

REFERENCES:
- [Derived] Hema-Ouangraoua S, Tranchot-Diallo J, Zongo I, Kabore NF, Nikiema F, Yerbanga RS, Tinto H, Chandramohan D, Ouedraogo GA, Greenwood B, Ouedraogo JB. Impact of mass administration of azithromycin as a preventive treatment on the prevalence and resistance of nasopharyngeal carriage of Staphylococcus aureus. PLoS One. 2021 Oct 13;16(10):e0257190. doi: 10.1371/journal.pone.0257190. eCollection 2021. PMID 34644317
- [Derived] Cairns ME, Sagara I, Zongo I, Kuepfer I, Thera I, Nikiema F, Diarra M, Yerbanga SR, Barry A, Tapily A, Coumare S, Milligan P, Tinto H, Ouedraogo JB, Chandramohan D, Greenwood B, Djimde A, Dicko A. Evaluation of seasonal malaria chemoprevention in two areas of intense seasonal malaria transmission: Secondary analysis of a household-randomised, placebo-controlled trial in Hounde District, Burkina Faso and Bougouni District, Mali. PLoS Med. 2020 Aug 21;17(8):e1003214. doi: 10.1371/journal.pmed.1003214. eCollection 2020 Aug. PMID 32822362
- [Derived] Chandramohan D, Dicko A, Zongo I, Sagara I, Cairns M, Kuepfer I, Diarra M, Barry A, Tapily A, Nikiema F, Yerbanga S, Coumare S, Thera I, Traore A, Milligan P, Tinto H, Doumbo O, Ouedraogo JB, Greenwood B. Effect of Adding Azithromycin to Seasonal Malaria Chemoprevention. N Engl J Med. 2019 Jun 6;380(23):2197-2206. doi: 10.1056/NEJMoa1811400. Epub 2019 Jan 30. PMID 30699301